CLINICAL TRIAL: NCT02530372
Title: Feasibility of the UriCap-F for Urine Collection in Hospitalized Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: G.R. Dome Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GRD-01F
Record Dates: First submitted 2015-08-16; First posted 2015-08-21 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UriCap-F (Experimental): The UriCap-F is an FDA cleared Class I device intended for urinary management in women.
  The device is comprised of a multiple use unit and a single use unit. The multiple use unit is intended to be reused by the same patient for up to 30 days. It is removed every 24 hours, rinsed under running water, dried and re-applied.
  The UriCap is held in position by means of a single-use medically approved adhesive tape.
  Interventions: Device: UriCap-F

INTERVENTIONS:
Device: UriCap-F — non-invasive urine collection device for women

SUMMARY:
The study will evaluate safety and effectiveness of the UriCap-F, a non-invasive urine collection device for women, in hospitalized patients who would otherwise be treated with an indwelling catheter, pads or diapers.

DETAILED DESCRIPTION:
Following various disease conditions such as trauma, orthopaedic surgery, and infections etc., patients may be bedridden and unable to void in a bedpan or to make their way to the toilet. For lack of a better solution for urinary management, indwelling catheter and diaper use is common in hospitalized patients. There is no externally applied urine collection device on the market today for women. In such situations an indwelling catheter is often placed to relieve patients while they are incapacitated, despite lack of urinary retention. Indwelling catheters, although effective, are associated with discomfort, pain, and urinary tract infections. In other cases diapers or absorbent pads may be used. These may be associated with skin irritation and infection.

The study will evaluate the UriCap-F, non-invasive urine collection devices for women, in hospitalized patients who are able to void or who are incontinent of urine

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years old
* Empties the bladder completely on voiding
* A clinical indication for an indwelling catheter, use of pads or diapers
* Patient has signed an informed consent form, is cooperative and willing to complete all study procedures
* Absence of localized disease at the site of device application - vaginal discharge, itching, inflammation or skin condition
* Agrees to genital hair removal.

Exclusion Criteria:

* Pregnant or breastfeeding
* Menstruation at time of enrolment
* Known allergy to silicon
* Dysuria
* Urinary retention - Post-void residual urine more than 300cc
* Hematuria or pyuria (turbidity) on visual inspection, according to investigator judgement.
* Diagnosed with acute renal failure according, to investigator judgement.
* Serious or unstable psychological condition (e.g., eating disorders, clinical depression, anxiety, emotionally labile) which, in the opinion of the Investigator, would compromise the patient's well-being or successful participation in the study
* Participating in another clinical study.
* Financial interest in the Sponsor Company or a competitor company by patient or a family member

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Device Events | 1-30 days
Use Safety as demonstrated by System Usability Score assessed by healthcare providers | 1 week
Effectiveness of the device to collect urine | 1-30 days
  Multiple variables will be assessed and their measurements aggregated to arrive at a number of events reported:
  * Leakage
  * Pooling of urine in the tubing
  * Tubing disconnections
  * Adhesive tape disconnections
  * Need for repositioning of device
  * Device malfunctions
Patient satisfaction in device use | 1-30 days
  Overall treatment satisfaction will be assessed by means of a "Treatment Satisfaction Questionnaire" administered at termination of device use.
Healthcare provider (HCP) satisfaction | up to 60 days
  Treatment satisfaction will be assessed by means of a "Treatment Satisfaction Questionnaire" administered after termination of all study patients
Patient Comfort | 1-30 days
  Comfort will be assessed by means of the "Universal Pain Assessment Scale" of 1-10, At every device application, every removal, and when patient complains of discomfort or pain.

SECONDARY OUTCOMES:
Effectiveness of defined device cleaning procedure for reuse | 1-30 days
  The reusable part will be visually inspected after cleaning for suitability for reuse. Devices which exhibit any of the following properties will be discarded: color change, residual soiling, loss of mechanical integrity, torn or rough edges. Effectiveness of the cleaning procedure will be measured as the average number of days the device can be reused.
Leakage as a result of device movement | 1-30 days
  To evaluate the correlation between leakage and device repositioning data

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, MD, Principal Investigator — No affiliation